CLINICAL TRIAL: NCT02053779
Title: The Impact of a Single Dose of GnRH Agonist (Triptorelin 0,1 mg) at the Time of Implantation on the Reproductive Outcome in IVF Cycles Triggered by a GnRH Agonist Followed by a Small Bolus of HCG the Day of Oocyte Retrieval
Brief Title: GnRH Agonist Trigger and Modified Luteal Phase Support, Adding a Bolus of GnRHa at the Time of Implantation - a RCT
Acronym: GTMLPSGI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Ibn Rochd (Other)
Responsible Party: Principal Investigator, benmachiche abdelhamid, Dr benmachiche abdelhamid, private infertility centre, Ibn rochd, constantine, Algeria, Centre Hospitalier Universitaire Ibn Rochd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27111969
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Infertility
Keywords: GnRH agonist; GnRH antagonist; Luteal phase
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRH-agonist (Experimental): Experimental Arm: Triptorelin 0.1 mg
  Interventions: Drug: Triptorelin 0.1mg
- Control Arm (No Intervention): Control Arm: No intervention

INTERVENTIONS:
Drug: Triptorelin 0.1mg — Triptorelin 0.1 mg administered subcutaneously 6 days after ovum pick-up (OPU) in IVF/ICSI cycles triggered by triptorelin 0.2 mg followed by hCG 1500 iu the day of OPU.
  Other Names: Decapeptyl 0.1 mg
  Arms: GnRH-agonist

SUMMARY:
Purpose:The aim of this project is to prospectively determine whether a single dose of GnRH-agonist administered at the time of implantation increases or not the reproductive outcome in patients undergoing in vitro fertilization ( IVF)/ intracytoplasmatic sperm injection(ICSI) triggered by a GnRH-agonist followed by a small bolus of human chorionic gonadotropin (hCG 1500 IU) the day of oocyte retrieval.

Acronyms:

GnRH: gonadotropin-releasing hormone FSH: follicle stimulating hormone LH: luteinizing hormone HCG:human chorionic gonadotropin IVF:In vitro fertilization ICSI:intracytoplasmatic sperm injection OHSS:ovarian hyperstimulation syndrome OMEGA: oocyte maturation employing GnRH-agonist OPU: ovum pick up NaCl: sodium chloride

DETAILED DESCRIPTION:
It has been reported in previous publications that the ovarian hyperstimulation syndrome (OHSS) was eliminated when GnRH agonist was used to trigger ovulation and the delivery rate has improved after modified luteal support especially when a small bolus of hCG is used on the day of oocyte retrieval. (OMEGA/HCG 1500 IU).

However, a risk difference of 7% in delivery rates is still in favor of HCG trigger. Thus, further modifications in the luteal phase supplementation are required in order to optimise the reproductive outcome after GnRH-agonist triggering.

Recently, many papers showed, that independently of the GnRH analogue used to prevent the premature LH surge, the addition of GnRH-agonist during the luteal phase seems to be beneficial in terms of pregnancy. Nevertheless, their use in practice is not yet admitted because of controversial results in terms of efficacy and safety particularly on the conceptus.

ELIGIBILITY:
Inclusion Criteria:

* Female age < 40 years
* Baseline FSH and LH < 12 IU/l.
* Body Mass Index > 18 and < 35 kg/m2
* No uterine (fibroids, mullerian malformations), ovarian ( endometrioma) or adnexa (hydrosalpinx) abnormalities
* Patients with at least one embryo at transfer time

Exclusion Criteria:

* Very high risk of OHSS (> 30 follicles > 12 mm the day of ovulation triggering).
* Reduced ovarian reserve
* Fertilization failure
* Severe endocrinopathy
* Azoospermia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 328 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
implantation rate | 5 weeks after IVF/ICSI
  number of gestational sacs per number of embryos transferred

SECONDARY OUTCOMES:
chemical pregnancy | 2 weeks after IVF/ICSI
  confirmed by beta-hCG 14 days post embryo transfer
clinical pregnancy | 5 weeks after IVF/ICSI
  appearance of yolk sac with foetal heart beat at 7 weeks of gestation
live birth | 26 weeks after IVF/ICSI
  birth of baby beyond 28 weeks of gestation

OTHER OUTCOMES:
ovarian hyperstimulation syndrome OHSS | from date of triggering until 2 weeks after pregnancy test
  frequency of moderate to severe OHSS

CONTACTS AND LOCATIONS:
Overall Officials: Abdelhamid benmachiche, Doctor, Principal Investigator — Ibn roch infertility centre, cité boussouf, Constantine Algeria
Locations (1):
- Ibn Rochd Infertility Centre, Constantine, Algeria